CLINICAL TRIAL: NCT02762708
Title: The Effect of Bariatric Surgery on Metabolism, the Metabolome and the Microbiome in Patients With Type 2 Diabetes
Brief Title: The Effect of Bariatric Surgery on Metabolism, the Metabolome and Microbiome in Patients With Type 2 Diabetes
Acronym: Microbiome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Meera Shah, M.B., Ch.B., Assistant Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-000179
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: Bariatric Surgery; Weight loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Weight Loss | interventions — Gastric Bypass; Bariatric Surgery; Caloric Restriction; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Roux-en-Y Gastric Bypass (RYGB) (Active Comparator): Subjects between the ages of 20-65 years of age seen for weight management in the Nutrition Clinic at Mayo Clinic, who have been approved for RYGB.
  Interventions: Procedure: Roux-en-Y Gastric Bypass (RYGB)
- Caloric restriction (Sham Comparator): Subjects between the ages of 20-65 years of age, with diagnosis of Type 2 diabetes mellitus or impaired fasting glucose. Subjects will undergo caloric restriction alone to mimic weight loss seen after gastric bypass surgery.
  Interventions: Behavioral: Caloric Restriction
- Exendin-9,39 (Active Comparator): Four subjects who have undergone RYGB surgery will be studied 4 weeks after surgery. Subjects will be randomized to receive an infusion of Exendin-9,39 or normal saline.
  Interventions: Drug: Exendin-9,39
- Normal Saline (Placebo Comparator): Four subjects who have undergone RYGB surgery will be studied 4 weeks after surgery. Subjects will be randomized to receive an infusion of Exendin-9,39 or normal saline.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass (RYGB) — Subjects will be studied prior to surgical intervention and 12 weeks post surgery. Subjects in surgical arm will start diet intervention after surgery. Follow up with dietary will be per standard of care following RYGB surgery.
  Other Names: Bariatric Surgery
  Arms: Roux-en-Y Gastric Bypass (RYGB)
Behavioral: Caloric Restriction — Subjects participating in caloric arm of this study will be asked to consume an identical diet that is controlled for caloric content and macronutrient composition. This is identical to that consumed by patient undergoing RYGB. Subjects in the caloric restriction arm will start the diet after the screening visit. Compliance will be monitored by alternating weekly meetings with a clinical psychologist and dietician.
  Arms: Caloric restriction
Drug: Exendin-9,39 — A subset of 4 subjects who have undergone RYGB surgery will be studied 4 weeks after surgery. Subjects will be randomized to receive an infusion of either Exendin-9,39 or normal saline. Exendin-9,39 blocks the action of specific hormones called "incretins" that are produced by the gut in health and in larger quantities after gastric bypass surgery.
  Arms: Exendin-9,39
Drug: Normal Saline — subset of 4 subjects who have undergone RYGB surgery will be studied 4 weeks after surgery. Subjects will be randomized to receive an infusion of either Exendin-9,39 or normal saline. Exendin-9,39 blocks the action of specific hormones called "incretins" that are produced by the gut in health and in larger quantities after gastric bypass surgery.
  Arms: Normal Saline

SUMMARY:
What are the benefits of undergoing Roux-en-Y gastric bypass surgery in improving type 2 diabetes outside of weight loss alone?

DETAILED DESCRIPTION:
Roux-en-y gastric bypass (RYGB) surgery leads to improvements in diabetes that occurs even before any significant weight loss is seen. What are the reasons for this? There is evidence in animals that changes in the composition of gut bacteria after RYGB may be responsible for improvements in how glucose is metabolized in the body. The study aims to correlate changes in the bacterial composition of the gut that occurs after surgery with improvements in glucose metabolism in people with type 2 diabetes. The investigators will do this by using validated methods to measure glucose metabolism and cutting edge technology to analyze the gut microbiome. A parallel group of patients with similar weight, height and age will undergo caloric restriction alone to mimic weight loss seen after RYGB. Participants will also undergo similar glucose metabolism studies and analysis of their gut bacterial composition. Thus, any difference seen between groups can be attributed to the surgery itself and may lead to identification of novel therapeutic options for diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-65 years of age.
* Seen at Mayo Clinic Nutrition Clinic and have received authorization for RYGB surgery.
* Type 2 Diabetes Mellitus or impaired fasting glucose with BMI >35 AND not interested in surgery but are interested in supervised caloric restriction.

Exclusion Criteria:

* Previous treatment with thiazolidinediones.
* Chronic antibiotic therapy.
* Active microvascular or macrovascular complications of diabetes.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03; Primary Completion 2018-01-06 (Actual); Study Completion 2018-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meera Shah, MBChB, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects that have undergone Roux-en-Y Gastric Bypass (RYGB) and were enrolled in the RYGB arm of trial period 'Study 1-RYGB vs Caloric Restriction', will be enrolled in the second trial period 'Study 2-Exendin (9,39) Amide study' 4 weeks postoperatively.
Period: Study 1 - RYGB vs Caloric Restriction
Arm/Group | Roux-en-Y Gastric Bypass (RYGB) | Caloric Restriction | Exendin-9,39 | Normal Saline
Started | 3 | 9 | 0 | 0
Completed | 3 | 7 | 0 | 0
Not Completed | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Period: Study 2 - Exendin (9,39) Amide Study
Arm/Group | Roux-en-Y Gastric Bypass (RYGB) | Caloric Restriction | Exendin-9,39 | Normal Saline
Started | 0 | 0 | 1 | 0
Completed | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 12 participants were enrolled in the overall study, which was comprised of two separate studies. One participant completed and was analyzed for both studies, resulting in a total of 13 participants analyzed for the Baseline Measures overall.
Groups:
- Total: Total of all reporting groups
Arm/Group | Roux-en-Y Gastric Bypass (RYGB) | Caloric Restriction | Exendin-9,39 | Normal Saline | Total
Number analyzed (Participants) | 3 | 9 | 1 | 0 | 13
Age, Categorical [Count of Participants; unit: Participants] — Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  Participants
    Study 1-RYGB vs Caloric Restriction: number analyzed (Participants) | 3 | 9 | 0 | 0 | 12
    Study 1-RYGB vs Caloric Restriction: <=18 years | 0 | 0 |  |  | 0
    Study 1-RYGB vs Caloric Restriction: Between 18 and 65 years | 3 | 9 |  |  | 12
    Study 1-RYGB vs Caloric Restriction: >=65 years | 0 | 0 |  |  | 0
    Study 2-Exendin (9,39) Amide Study: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1
    Study 2-Exendin (9,39) Amide Study: <=18 years |  |  | 0 |  | 0
    Study 2-Exendin (9,39) Amide Study: Between 18 and 65 years |  |  | 1 |  | 1
    Study 2-Exendin (9,39) Amide Study: >=65 years |  |  | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  Participants
    Study 1-RYGB vs Caloric Restriction: number analyzed (Participants) | 3 | 9 | 0 | 0 | 12
    Study 1-RYGB vs Caloric Restriction: Female | 2 | 6 |  | 0 | 8
    Study 1-RYGB vs Caloric Restriction: Male | 1 | 3 |  | 0 | 4
    Study 2-Exendin (9,39) Amide Study: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1
    Study 2-Exendin (9,39) Amide Study: Female |  |  | 1 |  | 1
    Study 2-Exendin (9,39) Amide Study: Male |  |  | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  Participants
    Study 1-RYGB vs Caloric Restriction: number analyzed (Participants) | 3 | 9 | 0 | 0 | 12
    Study 1-RYGB vs Caloric Restriction: Hispanic or Latino | 0 | 0 |  | 0 | 0
    Study 1-RYGB vs Caloric Restriction: Not Hispanic or Latino | 1 | 0 |  | 0 | 1
    Study 1-RYGB vs Caloric Restriction: Unknown or Not Reported | 2 | 9 |  | 0 | 11
    Study 2-Exendin (9,39) Amide Study: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1
    Study 2-Exendin (9,39) Amide Study: Hispanic or Latino |  |  | 0 |  | 0
    Study 2-Exendin (9,39) Amide Study: Not Hispanic or Latino |  |  | 1 |  | 1
    Study 2-Exendin (9,39) Amide Study: Unknown or Not Reported |  |  | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  Participants
    Study 1-RYGB vs Caloric Restriction: number analyzed (Participants) | 3 | 9 | 0 | 0 | 12
    Study 1-RYGB vs Caloric Restriction: American Indian or Alaska Native | 0 | 0 |  |  | 0
    Study 1-RYGB vs Caloric Restriction: Asian | 0 | 0 |  |  | 0
    Study 1-RYGB vs Caloric Restriction: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Study 1-RYGB vs Caloric Restriction: Black or African American | 0 | 0 |  |  | 0
    Study 1-RYGB vs Caloric Restriction: White | 3 | 9 |  |  | 12
    Study 1-RYGB vs Caloric Restriction: More than one race | 0 | 0 |  |  | 0
    Study 1-RYGB vs Caloric Restriction: Unknown or Not Reported | 0 | 0 |  |  | 0
    Study 2-Exendin (9,39) Amide Study: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1
    Study 2-Exendin (9,39) Amide Study: American Indian or Alaska Native |  |  | 0 |  | 0
    Study 2-Exendin (9,39) Amide Study: Asian |  |  | 0 |  | 0
    Study 2-Exendin (9,39) Amide Study: Native Hawaiian or Other Pacific Islander |  |  | 0 |  | 0
    Study 2-Exendin (9,39) Amide Study: Black or African American |  |  | 0 |  | 0
    Study 2-Exendin (9,39) Amide Study: White |  |  | 1 |  | 1
    Study 2-Exendin (9,39) Amide Study: More than one race |  |  | 0 |  | 0
    Study 2-Exendin (9,39) Amide Study: Unknown or Not Reported |  |  | 0 |  | 0
Region of Enrollment [Number; unit: participants] — Study 1-RYGB vs Caloric Restriction. Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  participants
    United States: number analyzed (Participants) | 3 | 9 | 0 | 0 | 12
    United States | 3 | 9 |  |  | 12
Region of Enrollment [Number; unit: participants] — Study 2-Exendin (9,39) Amide Study Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  participants
    United States: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1
    United States |  |  | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Fasting Glucose
Description: Blood sample taken after an overnight fast.
Time Frame: At baseline and 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Roux-en-Y Gastric Bypass (RYGB) | Caloric Restriction
Number analyzed (Participants) | 3 | 7
mmol/l
  Baseline | 6.1 (0.88) | 7.23 (0.98)
  12 weeks post intervention | 6.48 (1.7) | 5.89 (0.4)

2. Primary Outcome: Fasting Glucose
Description: Blood sample taken after an overnight fast.
Time Frame: 4 weeks post intervention
Population: The number of participants analyzed for the Normal Saline group at 4 weeks post intervention is zero because no subjects were enrolled in this arm.
Measure: Number; unit: mmol/l
Arm/Group | Exendin-9,39 | Normal Saline
Number analyzed (Participants) | 1 | 0
mmol/l | 4.75 |

3. Primary Outcome: Peak Glucose
Description: Blood sample taken after a meal.
Time Frame: baseline and 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Roux-en-Y Gastric Bypass (RYGB) | Caloric Restriction
Number analyzed (Participants) | 3 | 7
mmol/l
  Baseline | 11.35 (1.5) | 10.84 (1.39)
  12 weeks post intervention | 11.8 (3.25) | 10.04 (0.54)

4. Primary Outcome: Peak Glucose
Description: Blood sample taken after a meal.
Time Frame: 4 weeks post intervention
Population: as for outcome 2
Measure: Number; unit: mmol/l
Arm/Group | Exendin-9,39 | Normal Saline
Number analyzed (Participants) | 1 | 0
mmol/l | 8.15 |

5. Primary Outcome: Glucose AUC
Description: Area under the curve calculated from Oral Glucose Tolerance Test
Time Frame: 0 to 360 minutes post-meal at Baseline and 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: mmol/l.min
Arm/Group | Roux-en-Y Gastric Bypass (RYGB) | Caloric Restriction
Number analyzed (Participants) | 3 | 7
mmol/l.min
  Baseline | 2815 (223) | 2715 (375)
  12 weeks post intervention | 3146 (1186) | 2380 (139)

6. Primary Outcome: Changes in the Gut Microbiome Following RYGB or Caloric Restriction
Description: Stool sample collection for gut microbiome analysis
Time Frame: baseline and 12 weeks post intervention
Population: No participants samples were analyzed due to inability to obtain funding to proceed with gut microbiome analysis.
Arm/Group | Roux-en-Y Gastric Bypass (RYGB) | Caloric Restriction
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 12 weeks on all participants.
Description: Number of participants at risk for Serious Adverse Events, All-Cause Mortality and Other (Not Including Serious) Adverse Events is zero for the saline arm because no participants were enrolled in the saline arm of study 2- Exendin (9,39) Amide study period.
Arm/Group | Roux-en-Y Gastric Bypass (RYGB) | Caloric Restriction | Exendin-9,39 | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/9 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/9 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/9 | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Only one patient was enrolled in the trial period 'Study 2-Exendin (9,39) Amide study' 4 weeks post operatively. There were logistical challenges to recruiting patients 4 weeks post operatively as operation dates were not always known to the study team in time and patients did not feel well enough to come in for a study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT02762708/Prot_SAP_000.pdf